CLINICAL TRIAL: NCT03706651
Title: Assessment of Tele-expertise for the Interpretation of MRI Among Neonates With High Risk of Neurological Sequelae
Acronym: Matrix Neonat
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: TLM-MatrixNeonat
Record Dates: First submitted 2018-09-24; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Hypoxia, Brain
MeSH Terms: conditions — Hypoxia, Brain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed group, during Tele-expertise: Infants hospitalized in health facilities performing tele-expertise
  Interventions: Device: Infants hospitalized in health facilities performing Tele-expertise
- Exposed group, Prior Tele-expertise: Infants hospitalized in health facilities performing Tele-expertise prior implementation of Tele-expertise

INTERVENTIONS:
Device: Infants hospitalized in health facilities performing Tele-expertise
  Groups: Exposed group, during Tele-expertise

SUMMARY:
The purpose of the study is to determine whether tele-expertise would be more effective and more cost-effective for the Interpretation of MRI Among Neonates with high risk of neurological sequelae

ELIGIBILITY:
Inclusion Criteria:

* Less than 28 days of life
* Mandatory to have a medical advice in paediatric neuroradiology for interpretation of brain MRI

Exclusion Criteria:

* None

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants hospitalized in neonatology unit
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-01; Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Time between MRI and decision of intensive care continuation | 1 week after discharge
  A cerebral MRI for neonates, prescribed by the ICU team, will be performed, requiring a specialist advice. This advice is mandatory for ICU team to decide the intensive care continuation.

SECONDARY OUTCOMES:
Time between MRI and the specialist report | 1 week after discharge
Time between MRI and the discussions with the parents | 1 week after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Dion, MD, PhD, Principal Investigator — Centre de téléradiologie, Assistance Publique, Hôpitaux de Paris; Isabelle Durand-Zaleski, MD, PhD, Principal Investigator — DRCD URC Eco. Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Service de radiopédiatrie, Le Kremlin-Bicêtre
  - Service de Radiopédiatrie. Hôpital Trousseau, Paris
  - Service de radiopédiatrie. Hôpital Necker, Paris
  - Service de radiopédiatrie - Hôpital Robert Debré, Paris

REFERENCES:
- [Background] Larroque B, Ancel PY, Marret S, Marchand L, Andre M, Arnaud C, Pierrat V, Roze JC, Messer J, Thiriez G, Burguet A, Picaud JC, Breart G, Kaminski M; EPIPAGE Study group. Neurodevelopmental disabilities and special care of 5-year-old children born before 33 weeks of gestation (the EPIPAGE study): a longitudinal cohort study. Lancet. 2008 Mar 8;371(9615):813-20. doi: 10.1016/S0140-6736(08)60380-3. PMID 18328928
- [Background] Kidholm K, Ekeland AG, Jensen LK, Rasmussen J, Pedersen CD, Bowes A, Flottorp SA, Bech M. A model for assessment of telemedicine applications: mast. Int J Technol Assess Health Care. 2012 Jan;28(1):44-51. doi: 10.1017/S0266462311000638. PMID 22617736